CLINICAL TRIAL: NCT04462250
Title: Development of a Mobile Health App to Improve the Safe Use, Storage, and Disposal of Opioid Medications
Brief Title: Mobile Health (mHealth) App for Safe Opioid Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Rutgers, The State University of New Jersey (Other)
Responsible Party: Principal Investigator, Ann D. Bagchi, PhD, DNP, Assistant Professor, Rutgers, The State University of New Jersey
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Device Feasibility
Other Study IDs: Pro2020001699
Record Dates: First submitted 2020-07-01; First posted 2020-07-08 (Actual); Last update posted 2021-09-27 (Actual); Status verified 2021-09

CONDITIONS: Opioid Use

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Participants will enter all data using a numeric identifier assigned by a third-party recruiter
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Control (Active Comparator): Subjects will use the smartphone app to manage use of prescribed opioid medications to earn points but there will be no reward provided.
  Interventions: Device: Prescription Opioid Management App
- Contingency Management - Virtual Pet (Active Comparator): Subjects will use the smartphone app to manage use of prescribed opioid medications to earn points, which can be used in the care of a virtual pet.
  Interventions: Device: Prescription Opioid Management App
- Contingency Management - Monetary (Active Comparator): Subjects will use the smartphone app to manage use of prescribed opioid medications to earn points, which will be paid out at the end of the one-week trial in the form of a monetary reward.
  Interventions: Device: Prescription Opioid Management App

INTERVENTIONS:
Device: Prescription Opioid Management App — Smartphone application that provides education and reinforcement of safe opioid use, storage, and disposal

SUMMARY:
A key driver of the current opioid overdose epidemic is the misuse of legitimately prescribed opioid medications. Patient education through use of mobile technology may help to increase knowledge of appropriate use of opioid medications; however, knowledge does not always translate into behavior modification. Therefore, there is a need for more research into patient-facing technology that can increase both knowledge and behaviors consistent with appropriate opioid use. These needs have been amplified by the severe acute respiratory syndrome coronavirus-2 (COVID-19) pandemic, which has exposed healthcare disparities, heightened the risk for mental and behavioral health disorders, and dramatically increased reliance on telehealth technologies. It is critically important that telehealth solutions be accessible and user-friendly for all consumers, particularly members of underserved communities with limited digital health literacy. This feasibility study will develop a mobile health app to improve appropriate use of opioid medications among patients with a prescription to treat non-cancer pain. The study will use focus groups with consumers and providers to determine the content and features to be included in the app and will test the feasibility of implementing a contingency management approach (i.e., rewards system) with the app using a randomized control trial. The key outcome of interest is confirmation of the design and operating specifications of the app, including the use of contingency management. Secondary outcomes of interest are the overall rating of the app and an increase in knowledge among users regarding the safe use, storage, and disposal of opioid medications.

ELIGIBILITY:
Inclusion Criteria:

* Has current prescription for opioid medication
* Any ethnic group
* Served through the following programs of partnering organization: primary medical care, transgender medical care, HIV and sexually transmitted infection (STI) screening and counseling, LGBTQ services, pre-exposure prophylaxis and post exposure prophylaxis services, health education, clinical research, case management, psychosocial services, nutrition counseling, treatment adherence
* Owns an Android-base smartphone

Exclusion Criteria:

* Unable to provide informed consent
* Pregnant women
* Currently being treated for/history of mental health or substance use disorder

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-08-24 (Actual); Primary Completion 2022-02-28 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Device functionality | Assessed at the end of the one-week trial
  Confirmation that the app features work as intended based on user input

SECONDARY OUTCOMES:
Mobile App Rating Scale (MARS) | Data collected through app and telephone interviews at the end of the one-week trial
  Participants' assessment of functionality and utility of app with 19 items scored from 1 to 5 (overall score range 19 to 95) where higher scores indicate better app rating
Change in knowledge quiz score | Change in score as assessed at the end of the one-week trial
  Participants will show an increase in knowledge related to the safe used, storage, and disposal of opioid medications based on a 10-item, investigator created, pre/post quiz (total score range of 1 to 10) designed to address key educational components of the app

CONTACTS AND LOCATIONS:
Overall Officials: Ann D Bagchi, PhD,DNP, Principal Investigator — Rutgers, The State University of New Jersey
Locations (1):
- North Jersey Community Research Initiative, Newark, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data